CLINICAL TRIAL: NCT01348321
Title: Superior Efficacy of Azithromycin and Levamisole Versus of Azithromycin Alone in the Treatment of Inflammatory Acne Vulgaris: An Investigator Blind Randomized Clinical Trial on 169 Patients
Brief Title: Comparison of Efficacy of Azithromycin and Levamisole Versus of Azithromycin in in the Treatment of Acne
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ahvaz Jundishapur University of Medical Sciences (Other)
Responsible Party: Sima Rasaii, Jundishapur University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acne and levamisole; 126/د (Other: Ajums)
Record Dates: First submitted 2011-04-25; First posted 2011-05-05 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2008-10

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Levamisole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromicine plus levamisole (Experimental)
  Interventions: Drug: Levamisole
- Azithromicin (Experimental)
  Interventions: Drug: Levamisole

INTERVENTIONS:
Drug: Levamisole — Group 1: Azithromycin 500 mg per day, three days a week plus oral levamisole 150 mg per day, two days a week. Group 2: Azithromycin 500 mg per day, three days a week. The used medications were not revealed to their physician. A questionnaire was filled for every patient and photos were taken from lesions using a digital camera at first, second and final visit.

SUMMARY:
Different immunologic mechanisms contribute to development of inflammation in acne vulgaris and immunologic effect of levamisole has been demonstrated.

Objective: The aim of this study was to compare azithromycin and levamisole with azithromycin alone in the treatment of acne vulgaris.

DETAILED DESCRIPTION:
An investigator blind clinical randomized prospective two months study was designed. One hundred sixty nine acne patients presenting in our outpatients clinic were randomly allocated to two treatment groups: azithromycin and levamisole ( group 1 ) and azithromycin alone ( group 2 ) .One hundred forty eight patients completed the duration of the study and their clinical responses were evaluated and compared by using monthly photographic records .

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had at least 20 papules and/or pustules,
2. Patients with nodule and/or cyst disregarding the number of papules of pustules, were included the study. There was not any age limit

Exclusion Criteria:

1. were using any type of systemic treatment for their acne at the time of visit or during the last month;
2. had any hematological, renal or hepatic disease
3. were pregnant or lactating;
4. had drug-induced acne;
5. were using alcohol, anti-convulsants or anti-coagulants.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | one year
  A questionnaire was filled for every patient.For patients in both groups, lab tests were done at each visit.All adverse effect and the number of them were recorded and the patients who had side-effects or didn't follow the visits were excluded from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sima Rasaii, Dermtologist, Principal Investigator — Jundishapur University of Medical Sciences
Locations (1):
- Azadegan Street,Imam Hospital,Department of Dermatology, Ahvāz, Khoozestan, Iran

REFERENCES:
- [Background] Haneke E. [Levamisole treatment of acne fulminans (author's transl)]. Z Hautkr. 1981 Sep 1;56(17):1160-6. German. PMID 6457452
- [Result] Ansarin H, Savabynasab S, Behzadi AH, Sadigh N, Hasanloo J. Doxycycline plus levamisole: combination treatment for severe nodulocystic acne. J Drugs Dermatol. 2008 Aug;7(8):737-40. PMID 18720689
- [Derived] Rassai S, Mehri M, Yaghoobi R, Sina N, Mohebbipour A, Feily A. Superior efficacy of azithromycin and levamisole vs. azithromycin in the treatment of inflammatory acne vulgaris: an investigator blind randomized clinical trial on 169 patients. Int J Clin Pharmacol Ther. 2013 Jun;51(6):490-4. doi: 10.5414/CP201861. PMID 23547851